CLINICAL TRIAL: NCT06622343
Title: Risk Factor Analysis and Predictive Modeling for Necrotizing Skin Infections in Venomous Snakebite Patients: A Multicenter Retrospective Study
Brief Title: Predictive Modeling of Necrotizing Skin Infections in Snakebite Patients
Status: Completed | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Central People's Hospital of Zhanjiang (Other); Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Principal Investigator, Zhibin Xu, Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: KY20240521-001
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Necrotizing Skin Infections; Snakebite Envenomation
Keywords: Snakebite; Necrotizing Infection; Risk Factors; Predictive Modeling; Venomous Snakes; D-dimer; Snakebite Severity Score; Blood Glucose Levels
MeSH Terms: conditions — Snake Bites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — This study involved the collection of blood samples from patients upon hospital admission. The samples were used to measure key clinical markers such as blood glucose levels, D-dimer, C-reactive protein (CRP), white blood cell count (WBC), and other relevant biomarkers. These biospecimens were analyzed to identify potential predictors of necrotizing skin infections in patients with venomous snakebites. The samples were collected and processed according to standardized clinical protocols, but they were not retained for future genetic or DNA-based research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Necrotizing Skin Infections Group: This cohort includes patients who developed necrotizing skin infections following venomous snakebites. These patients were treated at three hospitals in Guangdong Province between January 2020 and April 2024. The study aims to identify key risk factors, including Snakebite Severity Score (SSS), blood glucose levels, and D-dimer levels, that are associated with the development of necrotizing skin infections in these patients.
  Interventions: Drug: Antivenom Serum; Procedure: Wound Debridement
- Non-Infection Group: This cohort includes patients who did not develop necrotizing skin infections after venomous snakebites. These patients were treated at the same three hospitals between January 2020 and April 2024. The cohort serves as a control group to compare against the infection group, helping to determine risk factors associated with necrotizing skin infections in snakebite patients.
  Interventions: Drug: Antivenom Serum; Procedure: Wound Debridement

INTERVENTIONS:
Drug: Antivenom Serum — Intravenous administration of 6000 IU of antivenom serum was given to patients envenomed by pit vipers. This treatment was based on Chinese guidelines for the management of snakebites. Additionally, patients received supportive treatments, including antibiotics to prevent infection, antihistamines for allergic reactions, and magnesium sulfate for localized swelling and pain relief.
Procedure: Wound Debridement — Patients who did not develop necrotizing skin infections received wound management, including multiple punctures using a three-edged needle for toxin drainage, along with standard wound care and debridement as necessary to prevent infection and promote healing.

SUMMARY:
This multicenter retrospective study aims to identify the risk factors associated with necrotizing skin infections following venomous snakebites and to develop a predictive model. Clinical data from 99 patients treated between January 2020 and April 2024 at three hospitals in Guangdong Province, China, were analyzed.

DETAILED DESCRIPTION:
Venomous snakebites are a significant public health issue, particularly in tropical and subtropical regions like southern China. Necrotizing skin infections are a severe but relatively rare complication of venomous snakebites, often resulting from delayed treatment and bacterial invasion. This study retrospectively analyzed clinical data from 99 patients with venomous snakebites treated at three hospitals in Guangdong Province between January 2020 and April 2024. The primary objective was to identify the major risk factors associated with the development of necrotizing skin infections and to build a predictive model to assist in clinical decision-making.

The study included male and female patients aged 14 years and older. Patients with incomplete medical records, long-term use of immunosuppressants, or underlying immunodeficiency diseases were excluded. Multivariate logistic regression identified the Snakebite Severity Score (SSS), blood glucose levels, and D-dimer levels as significant independent predictors of necrotizing infections.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of venomous snake bites confirmed according to major international clinical guidelines and expert consensus.
* Availability of complete case data.
* Provision of written informed consent by the patients or their legal guardians.

Exclusion Criteria:

* Age less than 14 years.
* Long-term use of immunosuppressants or corticosteroids.
* Presence of concurrent immunodeficiency diseases (e.g., HIV positive).
* Severe malnutrition.
* Incomplete medical records.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients (aged 18 years and older) who were treated for venomous snakebites at three hospitals in Guangdong Province. The population consists of both male and female patients with confirmed envenomation and sufficient medical records for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Necrotizing Skin Infections | 30 days from admission or until discharge.
  The primary outcome measure is the incidence of necrotizing skin infections among venomous snakebite patients within the study period. Necrotizing infections were identified based on clinical diagnostic criteria, including tissue necrosis, infection severity, and systemic symptoms.

SECONDARY OUTCOMES:
Hospital Length of Stay | From hospital admission until discharge, typically ranging between 1 and 30 days.
  The secondary outcome measure is the duration of hospitalization for patients with venomous snakebites, comparing those who developed necrotizing skin infections with those who did not.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong, China